CLINICAL TRIAL: NCT05176717
Title: A Double-Masked, Randomized, Controlled, Multiple-Dose Study to Evaluate the Efficacy, Safety and Tolerability of QR-421a in Subjects With Retinitis Pigmentosa (RP) Due to Mutations in Exon 13 of the USH2A Gene With Early to Moderate Vision Loss
Brief Title: Study to Evaluate the Efficacy Safety and Tolerability of QR-421a in Subjects With RP Due to Mutations in Exon 13 of the USH2A Gene With Early to Moderate Vision Loss (Celeste)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Laboratoires Thea (Industry)
Collaborators: Sepul Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PQ-421a-004; 2021-002728-19 (EudraCT Number)
Record Dates: First submitted 2021-11-23; First posted 2022-01-04 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Retinitis Pigmentosa; Usher Syndrome Type 2; Deaf Blind; Retinal Disease; Eye Diseases; Eye Diseases, Hereditary; Eye Disorders Congenital; Vision Disorders
Keywords: Retinitis Pigmentosa; USH2A; RP; exon 13; RNA therapies; antisense oligonucleotide; exon skipping; Celeste; IVT; mutations in exon 13 of the USH2A gene; NSRP; Intravitreal Injection; Non-Syndromic RP; Inherited Retinal Diseases; Usher Syndrome
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Eye Abnormalities; Vision Disorders | interventions — Intravitreal Injections

STUDY DESIGN:
Intervention Model Description: After primary endpoint is assessed at 12 months, subjects continue the same randomized treatment in the fellow eye. Subjects enrolled to sham treatment will be randomized to receive one of the two ultevursen doses in a parallel design fashion.
  Double-masked, randomized, controlled, multiple-dose study. Subjects will be randomized to one of three treatment groups:
  1. Group 1: QR-421a 180/60 µg (180 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter)
  2. Group 2: QR-421a 60/60 µg (60 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter; n = 27)
  3. Group 3: Sham-procedure (administered on Day 1, Month 3 and every 6 months thereafter; n = 27)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subject, site staff (study coordinator, imaging technician, etc) and Investigator will be completely masked. Physician performing IVT and post-IVT monitoring will know if subject is receiving sham or treatment, but will be masked to the dose level. Pharmacist is the only site staff that will be completely unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- QR-421a 180/60 µg (Experimental): 180 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter
  Interventions: Drug: QR-421a
- QR-421a 60/60 µg (Experimental): 60 µg loading dose administered on Day 1, 60 µg maintenance dose administered at Month 3 and every 6 months thereafter
  Interventions: Drug: QR-421a
- Sham-procedure (Sham Comparator): Sham-procedure (no experimental drug administered) on Day 1, Month 3 and every 6 months thereafter
  Interventions: Other: Sham-procedure

INTERVENTIONS:
Drug: QR-421a — RNA antisense oligonucleotide for intravitreal injection
  Other Names: RNA antisense oligonucleotide for intravitreal injection
  Arms: QR-421a 180/60 µg; QR-421a 60/60 µg
Other: Sham-procedure — Sham-procedure (no experimental drug administered)
  Arms: Sham-procedure

SUMMARY:
The purpose of this study is to evaluate the efficacy safety and tolerability of QR-421a administered via intravitreal injection (IVT) in subjects with Retinitis Pigmentosa (RP) due to mutations in exon 13 of the USH2A gene with early to moderate vision loss.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy safety and tolerability of QR-421a administered via intravitreal injection (IVT) in subjects with Retinitis Pigmentosa (RP) due to mutations in exon 13 of the USH2A gene with early to moderate vision loss.

The below dose levels of QR-421a will be evaluated with the loading dose administered at Day 1 and maintenance dose administered at Month 3 and every 6 months thereafter:

1. Loading dose of 180 μg, maintenance dose of 60 μg
2. Loading dose of 60 μg, maintenance dose of 60 μg

Dose levels will include subjects randomized to sham-procedure or treatment with QR-421a. After the study eye has been treated for at least 12 months, treatment of the fellow eye and cross-over of subjects assigned to sham-procedure may be initiated in eligible eyes based on assessment of benefit-risk.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age OR a minor (12 to < 18 years) with permission from a parent or legal guardian.
2. An adult willing to comply with the protocol, follow study instructions, attend study visits as required and willing and able to complete all study assessments. OR A minor able to complete all study assessments and comply with the protocol and has a parent or caregiver willing and able to follow study instructions, and attend study visits with the subject as required.
3. Clinical presentation consistent with RP with Usher syndrome type 2 or nonsyndromic form of RP (NSRP), based on ophthalmic, audiologic, and vestibular examinations.
4. A molecular diagnosis of homozygosity or compound heterozygosity for 1 or more pathogenic exon 13 mutations in the USH2A gene, based on genetic analysis at screening.
5. BCVA better than ≥69 letters (approximate Snellen equivalent 20/40) in the study eye, using the best BCVA reading at Screening.
6. Impairment of Visual Field (VF) in the opinion of the Investigator as determined by perimetry, with a continuous area of central field greater than or equal to 10 degrees diameter in each meridian as measured by a size V4e target, and a mean defect of ≥ 10 dB, in the study eye.
7. Clearly visible and measurable ellipsoid zone (EZ) width and/or area on SDOCT, per investigator judgement.
8. No limitations to SD-OCT image collection that would prevent high quality, reliable images from being obtained in both eyes, as determined by the Investigator.
9. Reliable Best Corrected Visual Acuity (BCVA), perimetry, and other measurements in both eyes, as described in the Study Reference Manual and Imaging Manual and determined by the Investigator.
10. No visually significant ocular media opacities and adequate pupillary dilation to permit good quality retinal imaging, as assessed by the Investigator.

Exclusion Criteria:

1. Presence of additional non-exon 13 USH2A pathogenic mutation(s) on the USH2A allele carrying the exon 13 mutation in subjects who have monoallelic exon-13 mutations.
2. Presence of non-exon 13 USH2A pathogenic mutation(s) on both USH2A alleles in subjects who have biallelic exon 13 mutations.
3. Presence of pathogenic mutations in genes (other than the USH2A gene) associated with Usher syndrome Type 2 or NSRP, or other inherited retinal degenerative diseases or syndromes. Note: The confirmed presence of homozygous or compound heterozygous known disease-causing mutations in other genes involved in recessive retinal dystrophies (RD), or the confirmed presence of known disease-causing mutations in genes involved in dominant or X-linked retinal dystrophies is exclusionary.
4. Presence of any significant ocular or non-ocular disease/disorder (or medication and/or laboratory test abnormalities) which, in the opinion of the Investigator and with concurrence of the Medical Monitor, may either put the subject at risk because of participation in the study, may influence the results of the study, or the subject's ability to participate in the study. This includes but is not limited to a subject who has uncontrolled cystoid macular edema (CME) in the study eye. CME is permissible if stable for 3 months (with or without treatment). Past CME is permissible if resolved for more than 1 month.
5. History or presence of ocular herpetic diseases (including herpes simplex virus, varicella zoster or cytomegalovirus) in either eye.
6. Presence of any active ocular infection in either eye.
7. Presence of any of the following lens opacities in the study eye: cortical opacity ≥ +2, posterior subcapsular opacity ≥ +2, or a nuclear sclerosis ≥ +2, and which are: 1) clinically significant in the opinion of the Investigator, 2) would adequately prevent clinical and photographic evaluation of the retina.
8. History of amblyopia in the study eye that resulted in significant vision loss, in the opinion of the Investigator.
9. Receipt within 3 months prior to Screening of any intraocular or periocular surgery (including refractive surgery), or an IVT injection other or planned intraocular surgery or procedure during the course of the study.
10. Current treatment or treatment within the past 12 months with therapies known to influence the immune system (including but not limited to steroid implants, cytostatics, interferons, tumor necrosis factor (TNF)-binding proteins, drugs acting on immunophilins, or antibodies with known impact on the immune system). Subjects that have been treated with systemic steroids within the past 12 months or that require intermittent use of topical steroids may be considered for inclusion following approval by the Medical Monitor.
11. A history of glaucoma or an IOP greater than 24 mmHg in either eye that is not controlled with medication or surgery.
12. Use of any investigational drug or device within 90 days or 5 half-lives preceding the first dose of study medication, whichever is longer, or plans to participate in another study of an investigational drug or device during the course of the study.
13. Any prior treatment with genetic or stem-cell therapy for ocular or non-ocular disease.
14. History of malignancy within 2 years prior to Screening, except adequately treated squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
15. Known hypersensitivity to antisense oligonucleotides or any constituents of the injection.
16. Pregnant and breastfeeding subjects. Females of childbearing potential and males must comply with using highly effective methods of contraception as defined in the protocol. Women of non-childbearing potential may be included without the use of adequate birth control.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sepul Bio Chief Medical Officer, Study Director — Sepul Bio; Sepul Bio Clinical Operations Director, Study Director — Sepul Bio
Locations (3):
- United States (2):
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Wisconsin - Madison, Madison, Wisconsin
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QR-421a 180/60 µg | QR-421a 60/60 µg | Sham-procedure
Started | 1 | 2 | 2
Completed | 0 | 0 | 0
Not Completed | 1 | 2 | 2
Not completed — Sponsor Decision | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QR-421a 180/60 µg | QR-421a 60/60 µg | Sham-procedure | Total
Number analyzed (Participants) | 1 | 2 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13 | 34 (11.3) | 27 (19.8) | 27 (14.3)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: Adult (>= 18 years) | 0 | 2 | 1 | 3
  Age Group: Pediatric (<18 years) | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Genotype - Heterozygous [Count of Participants; unit: Participants] | 1 | 2 | 2 | 5
Phenotype [Count of Participants; unit: Participants]
  Syndromic | 1 | 1 | 1 | 3
  Non-Syndromic | 0 | 1 | 1 | 2
Baseline Best Corrected Visual Acuity (BCVA) - Treated Eye [Mean (Standard Deviation); unit: Letters] — Baseline Best Corrected Visual Acuity (BCVA) is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) vision chart after mandatory manifest refraction.
  Letters | 73 | 78.5 (0.7) | 74 (1.4) | 75.6 (2.8)
Baseline Best Corrected Visual Acuity (BCVA) - Contralateral Eye [Mean (Standard Deviation); unit: Letters] — Baseline Best Corrected Visual Acuity (BCVA) is assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) vision chart after mandatory manifest refraction.
  Letters | 74.0 | 83.5 (6.4) | 74 (8.5) | 77.8 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sensitivity
Description: Change from baseline in mean sensitivity (based on static perimetry) at 12 months of treatment versus sham-procedure
Time Frame: 12 months
Population: Study prematurely terminated due to sponsor decision for reasons unrelated to safety
Arm/Group | QR-421a 180/60 µg | QR-421a 60/60 µg | Sham-procedure
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Ellipzoid Zone Area (EZ) as Measured by Spectral Domain Optical Coherence Tomography SD-OCT
Description: Ellipzoid Zone area (EZ) as measured by Spectral Domain optical coherence tomography SD-OCT
Time Frame: 27 months
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: Change from baseline in Best Corrected Visual Acuity (BCVA)
Time Frame: 27 months
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Spectral Domain Optical Coherence Tomography (SD-OCT) (Other Measures)
Description: Change from baseline in Spectral domain optical coherence tomography (SD-OCT) (other measures)
Time Frame: 27 months
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Low Luminance Visual Acuity (LLVA)
Description: Change from baseline in Low Luminance Visual Acuity (LLVA) using the ETDRS vision chart
Time Frame: 27 months
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Other Measures of Static Perimetry
Description: Change from baseline in other measures of static perimetry on the Octopus 900 as assessed by a central reading center
Time Frame: 27 months
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in Full-field Stimulus Threshold (FST)
Description: Change from baseline in Full-field Stimulus Threshold (FST) on the Diagnosys FST as assessed by a central reading center
Time Frame: 27 months
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in PRO Measure as Assessed by Michigan Retinal Degeneration Questionnaire (MRDQ)
Description: Change from baseline in PRO measure as assessed by Michigan Retinal Degeneration Questionnaire (MRDQ)
Time Frame: 27 months
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in PRO Measures as Assessed by Patient Global Impressions of Severity (PGI-S)
Description: Change from baseline in PRO measures as assessed by Patient Global Impressions of Severity (PGI-S)
Time Frame: 27 months
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in PRO Measures as Assessed by Patient Global Impressions of Change (PGI-C)
Description: Change from baseline in PRO measures as assessed by Patient Global Impressions of Change (PGI-C)
Time Frame: 27 months
Reporting Status: Not Posted

11. Secondary Outcome: Ocular and Non-ocular Adverse Events (AEs)
Description: Ocular and non-ocular adverse events (AEs)
Time Frame: 27 months
Reporting Status: Not Posted

12. Secondary Outcome: Cmax of QR-421a in Serum
Description: Maximum concentration (Cmax) of QR-421a in serum
Time Frame: 27 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change From Baseline in Mobility Course Score
Description: Change from baseline in mobility course score
Time Frame: 27 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 months, 18 days - Study was terminated prematurely, therefore follow-up maximum range is from the Screening visit to the End of Study visit, for each participant.
Description: Any event/condition noted once the subject receives their first dose of study drug until the End of study visit (30 days +/- 14 days post last dose of study drug).
Arm/Group | QR-421a 180/60 µg | QR-421a 60/60 µg | Sham-procedure
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QR-421a 180/60 µg (N=1) | QR-421a 60/60 µg (N=2) | Sham-procedure (N=2)
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Retinal pigmentation (Eye disorders) | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study prematurely terminated due to sponsor decision for reasons unrelated to safety

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution shall be free to publish, present, or use any Data and results arising out of its performance of the protocol. At least 30 days prior to submission for publication, institution shall submit to Sponsor for review and comment any proposed oral or written publication. Institution will consider any such comments in good faith but is under no obligation to incorporate Sponsor's suggestions. The review period for abstracts or poster presentations shall be 30 days.

DOCUMENTS (2):
  • Study Protocol (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT05176717/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT05176717/SAP_001.pdf